CLINICAL TRIAL: NCT04480216
Title: MAgnetic Gastrointestinal Universal Septotome: a Safety and Feasibility Study
Brief Title: MAgnetic Gastrointestinal Universal Septotome: a Safety and Feasibility Study (MAGUS)
Acronym: MAGUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P2019/643
Record Dates: First submitted 2020-02-27; First posted 2020-07-21 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-12

CONDITIONS: Diverticulum, Esophageal; Post Gastric Surgery Syndrome
MeSH Terms: conditions — Diverticulum, Esophageal; Dumping Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MAGUS — An upper endoscopy will be performed with the use of fluoroscopy. The MAGUS will be placed under fluoroscopy. The good positioning and the absence of any complications will be confirmed by gastroscopy.
  An injection of contrast agent will be done to be sure of the correct positioning and that no complications was happened.
  The patient will be kept overnight, with liquid food for 2 and mashed food up to 7 days post procedure

SUMMARY:
A novel magnetic device, called MAgnetic Gastrointestinal Universal Septotome (MAGUS) was designed to improve the Treatment of diverticulum of the esophagus, Pseudo-diverticulum of the upper GI tract, Candy cane syndrome This study aims to evaluating the safety of the feasability of this new device.

DETAILED DESCRIPTION:
In this study, the investigators aim at treating different pathological conditions, resulting in the appearance of a septum separating a healthy pathway and a pathological pouch. Food then stagnate in this pouch and results in different symptoms including dysphagia, pain and/or regurgitation or postprandial dysrhythmia.

Esophageal diverticula consists in the apparition of a pouch (diverticulum) alongside the esophagus. Some post-surgical conditions can result in the appearance of pseudo-diverticulum or afferent limb that transforms into a large pouch. One example is the candy cane syndrome, being an afferent loop syndrome post gastrectomy or post Roux-en-Y Gastric Bypass, were the afferent limb becomes a structure similar to a large diverticulum.

All those pathological conditions could be solved by the marsupialization of those (pseudo-)diverticulum. For several years, Zenker's diverticula (pharyngo-esophageal diverticulum) have been treated endoscopically using this technique, providing good clinical results. However, it is difficult to go further than the pharynx with this technique, since it needs specific semi-rigid tools and a stable cutting position. Hence, for further septa of the GI tract, the classic treatment is thoracoscopy and thoracotomy or laparoscopy and laparotomy, depending on the site. Those highly invasive procedures have a significant mortality and morbidity rate respectively of more than 5% and 20% and are liked to different complications including abdominal pain, port site wound infections, intraabdominal collection or anastomosis ulcer.

The MAGUS device consists of a flexible catheter preloaded with a magnetic device, made of two magnets linked by a wire. Each magnet is attached to the catheter and can be dropped separately from this catheter. The magnetic device aims to create an anastomosis by means of compression, using magnetic force and a retractable wire pulling system. For a given septum, the magnets are placed on either sides of the bottom of it. The retractable wire goes then from one another, passing on top of the septum. Both creates compression necrosis. This process induces eventually a cutting of the septum.

Once the cutting is performed, the magnets migrate and are expelled through natural ways.

The MAGUS device is an endoscopic procedure. Above standard of care monitoring, safety assessment of the procedure and device performance decreases the risk and unforeseen events.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Patient has got evaluable symptoms (dysphagia, regurgitation, pain, weight loss, halitosis or others) associated with one of the following pathology:

  1. Diverticulum of the esophagus;
  2. A pseudo-diverticulum of the upper GI tract;
  3. Candy cane syndrome;
* Willing and able to comply with the study procedures and provide written informed consent to participate in the study.

Exclusion Criteria:

* Refractory stenosis of the UGI proximal to the septum;
* Septum height smaller than 2,5 cm or higher than 6 cm (check through CT scan, Barium Swallow or other imaging method);
* Coagulation disorders;
* Previous implantation of a magnetic-sensitive medical device (including active electronic implant, metallic stent, …);
* Dysphagia related to motility disorder;
* Planned MRI in the following month (30 days) of intervention.
* Concurrent medical condition that would affect the investigator's ability to evaluate the patient's condition or could compromise patient safety;
* Patient went through a surgery less than 8 weeks before implantation of the magnets;
* Currently enrolled in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-02-19 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Technical magnet placement success | Day 0
  ability to deploy the MAGUS in satisfactory position across the septum (YES/NO)
Type of evacuation of the device | During 28 Days post-placement
  natural or endoscopic
Incidence of all adverse event | During 30 days post-placement
  SAE during device placement

SECONDARY OUTCOMES:
Number and type of AE after placement | During 3 month post placement
Patient's report of pain: visual analog scale | Before treatment - Day 1 - Day 14 - Day 28 - Month 3
  scored by a visual analog scale from 0 to 10 (0=no pain)
Number of unplanified interventions | During 3 months post-placement
Change of Eckardt and dysphagia score or GERD HRQL score | Before treatment - Day 1 - Day 14 - Day 28 - Month 3
Patient's satisfaction with the therapy: visual analogue scale | Day 14 - Day 28 - Month 3
  scored by a visual analogue scale from 0 to 10 (10= fully satisfied)
Emptying rate of the diverticular structure | Month 3
Difference of height of the septum cut before and after the treatment | Month 3
Change of SF12 quality of life score | Before treatment - Month 3

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Erasme, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rio-Tinto R, Huberland F, Van Ouytsel P, Delattre C, Dugardeyn S, Cauche N, Delchambre A, Deviere J, Blero D. Magnet and wire remodeling for the treatment of candy cane syndrome: first case series of a new approach (with video). Gastrointest Endosc. 2022 Jun;95(6):1247-1253. doi: 10.1016/j.gie.2021.12.027. Epub 2022 Jan 1. PMID 34979115
- [Derived] Huberland F, Rio-Tinto R, Cauche N, Dugardeyn S, Delattre C, Sandersen C, Rocq L, van Ouytsel P, Delchambre A, Deviere J, Blero D. Magnets and a self-retractable wire for endoscopic septotomies: from concept to first-in-human use. Endoscopy. 2022 Jun;54(6):574-579. doi: 10.1055/a-1554-0976. Epub 2021 Oct 29. PMID 34282579